CLINICAL TRIAL: NCT05447546
Title: A Phase 1, Single-Center, Randomized, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HT-6184 in Healthy Human Subjects
Brief Title: Study to Evaluate HT-6184 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halia Therapeutics, Inc. (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HT-6184-NHV-001
Record Dates: First submitted 2022-05-19; First posted 2022-07-07 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Normal Healthy Subjects

STUDY DESIGN:
Intervention Model Description: SAD portion in 4 cohorts, with 8 subjects in each cohort, 4 ascending single doses, MAD portion in 4 cohorts, with 8 subjects in each cohort, 4 multiple ascending doses.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- 1 mg HT-6184 QD (Active Comparator): Cohort 1 - 6 subjects x 1 mg HT-6184 QD on Day 1
  Interventions: Drug: HT-6184
- 1 mg Placebo QD (Placebo Comparator): Cohort 1 - 2 subjects x placebo, QD on Day 1
  Interventions: Drug: HT-6184 Placebo
- 2 mg HT-6184 QD (Active Comparator): Cohort 2 - 6 subjects x 2 mg HT-6184 QD on Day 1
  Interventions: Drug: HT-6184
- 2 mg Placebo QD (Placebo Comparator): Cohort 2 - 2 subjects x placebo, QD on Day 1
  Interventions: Drug: HT-6184 Placebo
- 3 mg HT-6184 QD (Active Comparator): Cohort 3 - 6 subjects x 3 mg HT-6184 QD on Day 1
  Interventions: Drug: HT-6184
- 3 mg Placebo QD (Placebo Comparator): Cohort 3 - 2 subjects x placebo, QD on Day 1
  Interventions: Drug: HT-6184 Placebo
- 4 mg HT-6184 QD (Active Comparator): Cohort 4 - 6 subjects x 4 mg HT-6184 QD on Day 1
  Interventions: Drug: HT-6184
- 4 mg Placebo QD (Placebo Comparator): Cohort 4 - 2 subjects x placebo, QD on Day 1
  Interventions: Drug: HT-6184 Placebo
- 1 mg HT-6184 QD x 2 weeks (Active Comparator): Cohort 5 - 6 subjects x 1 mg HT-6184 QD on Day 1-5, 8-12
  Interventions: Drug: HT-6184
- 1 mg Placebo QD x 2 weeks (Placebo Comparator): Cohort 5 - 2 subjects x 1 mg placebo, QD on Day 1-5, 8-12
  Interventions: Drug: HT-6184 Placebo
- 2 mg HT-6184 QD x 2 weeks (Active Comparator): Cohort 6 - 6 subjects x 2 mg HT-6184 QD on Day 1-5, 8-12
  Interventions: Drug: HT-6184
- 2 mg Placebo QD x 2 weeks (Placebo Comparator): Cohort 6 - 2 subjects x 2 mg placebo, QD on Day 1-5, 8-12
  Interventions: Drug: HT-6184 Placebo
- 3 mg HT-6184 QD x 2 weeks (Active Comparator): Cohort 7 - 6 subjects x 3 mg HT-6184 QD on Day 1-5, 8-12
  Interventions: Drug: HT-6184
- 3 mg Placebo QD x 2 weeks (Placebo Comparator): Cohort 7 - 2 subjects x 3 mg placebo, QD on Day 1-5, 8-12
  Interventions: Drug: HT-6184 Placebo
- 4 mg HT-6184 QD x 2 weeks (Active Comparator): Cohort 8 - 6 subjects x 4 mg HT-6184 QD on Day 1-5, 8-12
  Interventions: Drug: HT-6184
- 4 mg Placebo QD x 2 weeks (Placebo Comparator): Cohort 8 - 2 subjects x 4 mg placebo, QD on Day 1-5, 8-12
  Interventions: Drug: HT-6184 Placebo

INTERVENTIONS:
Drug: HT-6184 — Oral capsule
  Arms: 1 mg HT-6184 QD; 1 mg HT-6184 QD x 2 weeks; 2 mg HT-6184 QD; 2 mg HT-6184 QD x 2 weeks; 3 mg HT-6184 QD; 3 mg HT-6184 QD x 2 weeks; 4 mg HT-6184 QD; 4 mg HT-6184 QD x 2 weeks
Drug: HT-6184 Placebo — Oral capsule
  Arms: 1 mg Placebo QD; 1 mg Placebo QD x 2 weeks; 2 mg Placebo QD; 2 mg Placebo QD x 2 weeks; 3 mg Placebo QD; 3 mg Placebo QD x 2 weeks; 4 mg Placebo QD; 4 mg Placebo QD x 2 weeks

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of HT-6184 when administered as single oral doses at escalating dose levels in healthy volunteer subjects.

The secondary objectives of this study are to characterize the pharmacokinetics (PK) and pharmacodynamics (PD) of HT-6184. Results of the PD analyses will be used to determine the minimal biologically effective dose (MBED): the lowest dose that achieves >70% target inhibition compared to unstimulated vehicle controls over 24 hours in 4 of 6 treated volunteers.

DETAILED DESCRIPTION:
This is a phase 1, randomized, placebo-controlled, single-center, single and multiple ascending dose study designed to evaluate the safety, tolerability, PK, and PD of HT-6184.

Each cohort in the study will be comprised of 8 subjects, 6 subjects will receive HT-6184 and 2 subjects will receive placebo. A dose range of 1 mg - 4 mg HT-6184 will be explored in the SAD and MAD escalation cohorts in adult healthy volunteer subjects. Safety and PK data from the 8 completed cohorts will be reviewed.

For the SAD portion subjects will be divided into 4 cohorts of 8 subjects in each cohort. Four (4) ascending single doses (1 dose level per cohort) will be investigated.

Subjects will be screened for eligibility to participate in the study up to 26 days (Day -28) prior to admission to the study center on Day -2. Eligible subjects will be admitted to the study center on Day -2 and will be discharged on Day 2 after all scheduled assessments have been completed. Following discharge, subjects will return to the study center for follow-up visits on Day 7 and receive a follow-up phone call on Day 30.

A modified Fibonacci escalation schedule starting at 1 mg, (escalating by 100%) 2 mg, (escalating by 50%) 3 mg, and (escalating by 33%) 4 mg. The study will have an ongoing assessment of all available safety, tolerability, and concentration data prior to initiation of the next cohort.

For the MAD portion subjects will be divided into 4 cohorts of 8 subjects in each cohort. Four (4) ascending multiple doses (1 dose level per cohort) will be investigated.

Subjects will be screened for eligibility to participate in the study up to 26 days (Day -28) prior to admission to the study center on Day -2. Eligible subjects will be admitted to the study center on Day -2 and will be discharged on Day 13 after all scheduled assessments have been completed. Following discharge, subjects will return to the study center for a follow-up visit on Day 21 and receive a follow-up phone call on Day 42.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, between 18 and 65 years of age (inclusive) at Screening;
2. Has a body mass index (BMI) between 18.0 and 32.0 kg/m2 (inclusive) at Screening
3. Is in good general health, as determined by the Investigator, without clinically significant medical history;
4. Normal physical examination, 12-lead electrocardiogram (ECG), and vital signs, as determined by the Investigator;
5. Clinical laboratory values within the normal limits as defined by the clinical laboratory reference range;
6. Female partners of male participants of childbearing potential, and female participants of childbearing potential must agree to use a highly effective method of contraception prior to study entry, for the duration of study participation, and a minimum of 30 days after the last dose. Highly effective forms of contraception include the following:

   * Established use (i.e., at least 30 days prior to enrollment) of combined (estrogen and progestogen containing) oral, intravaginal or transdermal hormonal contraception associated with inhibition of ovulation,
   * Established use (i.e., at least 30 days prior to enrollment) progestogen-only oral, injectable or implantable hormonal contraception associated with inhibition of ovulation,
   * Established use (i.e., at least 30 days prior to enrollment) of an intrauterine device (IUD) or intrauterine hormone-releasing system (IUS),
   * bilateral tubal occlusion,
   * vasectomized partner, provided that partner is the sole sexual partner of the female trial participant and that the vasectomized partner has received medical assessment of the surgical success,
   * sexual abstinence, defined as refraining from heterosexual intercourse during the study, when this is in line with the preferred and usual lifestyle of the subject.
7. In the case of a female of childbearing potential, has a negative serum pregnancy test (SPT) at Screening and Day -2 and is willing to submit to a SPT at the end of study (EOS);
8. Negative urine test for drugs of abuse and breath test for alcohol use at Screening and check-in (Day -2). The tests may be repeated once if necessary and deemed appropriate by the Investigator;
9. Agree to refrain from tobacco or nicotine containing products within 48 hours prior to Day 1 and during the periods when PK blood samples are collected;
10. Agree to refrain from alcohol consumption within 48 hours prior to Day 1 and during the periods when PK blood samples are collected;
11. Agree to refrain from caffeine (i.e., coffee, tea, caffeinated soda, chocolate) within 48 hours prior to Day 1 and during the periods when PK blood samples are collected;
12. Agree to refrain from grapefruit, Seville oranges, and pomelo containing products within 72 hours prior to Day 1 and during the periods when PK blood samples are collected; and
13. Read, understand, and sign an informed consent.

Exclusion Criteria:

1. A female who is pregnant, plans to become pregnant during the study, or is breastfeeding a child;
2. Any clinically significant central nervous system, cardiac, pulmonary, renal, gastrointestinal (GI), endocrinological, respiratory, or metabolic conditions (or history), or other pathological or physiological conditions, that might interfere with the study results in the investigator's opinion;
3. Any condition which, in the investigator's opinion, puts the participant at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study;
4. Immunization within 10 days of Day 1;
5. Anticipated need for surgery or hospitalization during the study;
6. Consumed alcohol within 48 hours prior to Day 1 or refuses to abstain from alcohol throughout the duration of the study;
7. History of heavy smoking (i.e., more than 10 cigarettes a day or the tobacco/nicotine equivalent) within 3 months of screening or refuses to abstain from tobacco or nicotine-containing products throughout the duration of the study;
8. Donation or loss of blood (excluding volume drawn at screening) of ≥ 450 mL within 3 months of Day 1;
9. Active or lifetime infection (e.g., negative test for human immunodeficiency virus (HIV) and hepatitis, and no history of tuberculosis and syphilis) or a history of severe infection during the 30 days prior to screening;
10. Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment;
11. Prior treatment with a NLRP3 inhibitor for any indication;
12. Is unwilling or unable to refrain from using prescription medications for 30 days prior to Day 1 or over the counter medications, herbal preparations, and supplements for 14 days prior to Day 1 (excluding permitted forms of contraception and occasional use of acetaminophen [up to 2 g in 24 hours]);
13. Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator;
14. Is currently participating in any clinical trial;
15. Has received any investigational drug(s) within 30 days or 5 half-lives, whichever is longer, prior to study Day 1;
16. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data; and/or
17. Inability of the participant (or legally authorized representative) to comprehend the informed consent form (ICF) or unwillingness to sign the ICF.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events administered as single oral doses at escalating dose levels in healthy volunteer subjects. | up to 6 weeks
  Safety and tolerability of HT-6184 as measured by subject incidence of treatment-related adverse events.
Incidence of abnormal laboratory test results | up to 6 weeks
  Safety and tolerability of HT-6184 as measured by subject incidence of treatment-related abnormal lab values.
Incidence of treatment-emergent clinically abnormal electrocardiogram (ECG) | up to 6 weeks
  Safety and tolerability of HT-6184 as measured by subject incidence of treatment-related abnormal ECG.
Incidence of treatment-emergent clinically abnormal physical exam | up to 6 weeks
  Safety and tolerability of HT-6184 as measured by subject incidence of treatment-related abnormal physical exam.

SECONDARY OUTCOMES:
Plasma maximum measured drug concentration (Cmax) | up to 6 weeks
  Cmax will be reported.
Time of maximum concentration (Tmax) | up to 6 weeks
  Tmax will be reported.
Area under the plasma concentration-time curve (AUC0-24) | up to 6 weeks
  Area under the plasma concentration-time curve from 0 until 24 hours post-dose will be reported.
Area under the plasma concentration-time curve (AUC0-last) | up to 6 weeks
  Area under the plasma concentration-time curve, from 0 to the last quantifiable timepoint will be reported.
Area under the plasma concentration-time curve (AUC0-inf) | up to 6 weeks
  Area under the plasma concentration-time curve, from 0 to infinity will be reported.
Plasma half-life (T½) | up to 6 weeks
  T½ will be reported.
Terminal elimination rate constant (kel) | up to 6 weeks
  Terminal elimination rate constant will be reported.
Apparent clearance (CL/F) | up to 6 weeks
  CL/F will be reported.
Apparent volume of distribution at steady state (Vss/F) | up to 6 weeks
  Vss/F will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jesson Yeh, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States